CLINICAL TRIAL: NCT02721108
Title: Mindfulness Meditation Using a Smart-phone Application for Women With Chronic Pelvic Pain
Brief Title: Mindfulness Meditation for Chronic Pelvic Pain Management
Acronym: MEMPHIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Headspace UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 010817QM; 10925965 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2015-09-28; First posted 2016-03-28 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-06

CONDITIONS: Chronic Pelvic Pain
Keywords: Mindfulness; Headspace; Psychological approaches; Progressive muscle relaxation
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness: Group A (Experimental): Using a 60-day mindfulness instruction meditation app: 60 days of 10 and 20 minute long app modules with a spoken guide to mindfulness meditation, to be used once a day, including modules on the basics of mindfulness and a module targeted to pain, which can re-revisited until the end of the study
  Interventions: Behavioral: Mindfulness meditation
- Relaxation: Group B (Active Comparator): Using comparison relaxation app with a series of non-meditative progressive muscle relaxation instructions: 60 days of 10 and 20 minute long app modules to be used once per day with spoken words and relaxing sounds, which can re-revisited until the end of the study
  Interventions: Behavioral: Relaxation app
- Treatment as usual: Group C (No Intervention): No app: treatment as usual (watch and wait, medication and/or surgery) to investigate if any app intervention makes a difference to wellbeing and to ascertain dropout rates for the full-scale trial in patients who perceive that they are getting no intervention.

INTERVENTIONS:
Behavioral: Mindfulness meditation — The meditation content is a structured and progressive course, layering in new techniques and concepts over successive sessions. The course was created and narrated by a former monk - Andy Puddicombe - drawing on a secularised version of the techniques he was taught over 10 years' experience in monasteries around the world. The first 30 days cover basic techniques, assuming no previous experience of meditation. The second 30 days focus specifically on the use of these techniques with respect to pain. The duration of individual sessions builds over time. Days 1-10 are 10 minutes in duration, days 11-20 are 15 minutes in duration, and days 21-60 are 20 minutes in duration.
  Arms: Mindfulness: Group A
Behavioral: Relaxation app — The Active Control group will use the same app, but the app will be configured so that they will hear a series of non-meditative progressive muscle relaxation instructions, also narrated by Andy Puddicombe. These sessions will be identical every day, except that their duration will increase to mirror the increasing duration of the meditation content being listened to by the Intervention group.
  Arms: Relaxation: Group B

SUMMARY:
Chronic pelvic pain (CPP) in women is common, painful and disabling and puts much strain on women's lives and the (National Health Service) NHS.

CPP may be related to internal organs, the nervous system or psychological factors and is often difficult to treat. Surgery and drugs have risks and side effects, are expensive and do not help all patients.

Psychological treatments have potential to improve CPP but are not consistently available. Mindfulness meditation teaches people to accept their sensations and emotions in the present moment. This can help to accept pain better, which enables patients to focus on daily activities and improve their quality of life. It has been shown to help in headache, back pain and depression. Usually mindfulness meditation is taught by attending courses for 8 weeks.

The investigators want to find out in a full-scale trial if mindfulness meditation, taught by using a smartphone app, can help CPP patients.

In preparation for this full-scale study the investigators will conduct the MEMPHIS study to answer the following questions:

* How many patients are willing to participate?
* How often they use the app?
* Reasons for not wanting to participate/not using the app -

  - Which health questionnaires are the most useful ones?
* How many patients will be required for the full-scale trial?

Patients will receive the usual treatment and be divided into three groups

* using a 60-day mindfulness meditation app,

  -- using comparison app with progressive muscle relaxation but no meditation
* no app

Patients will complete health questionnaires, may be asked to comment in a focus group and record pain, medication changes, surgery and emergency medical visits

DETAILED DESCRIPTION:
CPP affects up to 24% women worldwide accounts for 20% of UK gynaecological clinic referrals and has a considerable impact on patients' quality of life and their income. CPP costs the NHS € 3.3bn per year. Despite costly interventions CPP is often resistant to surgical and medical treatment. Multifactorial psychological and somatic causes require a multidimensional approach. Psychological and somatic causes require a multidimensional approach, which is not routinely offered in gynaecology clinics.

Randomized Control Trial (RCT-) evidence suggests that primary inclusion of psychological interventions may be superior to primary surgery. Although psychological treatment is provided across the NHS, mostly in the context of primary care Improving Access to Psychological

Therapies there are problems with capacity, waiting times and overall number of patients being able to access services. Alternatively, patient self-management (PSM) is now recognised as a tool empowering patients to cope better with their condition.

Mindfulness meditation is a potentially valuable PSM tool in CPP.

The investigators conducted a systematic search of literature (07/2013, updated 12/2013) and found no RCTs on mindfulness meditation in CPP. However, two small pilot trials, one in CPP and one in endometriosis patients with promising results.

The investigators decided to undertake a systematic review on the effect of mindfulness meditation and extend the search to other chronic pain conditions (e.g. back pain, headache, fibromyalgia and diabetic neuropathy) because previous systematic reviews had number of limitations, such as not reporting effect size. Two independent reviewers assessed the risk of bias systematically using Review Manager (RevMan) 5.2 software. Out of 472 citations 9 RCTs were finally included. Most studies were of moderate quality; sample sizes were generally small.

Mindfulness meditation had positive effects on depression in chronic pain patients (SMD -0.28; 95%CI -0.53, -0.03; p = 0.03). A trend in reduction of anxiety and affective pain and a trend towards better QUOL, especially the mental health component and better pain acceptance was observed. Only one of the included studies reported the important measure of pain acceptance. If a larger sample size had been available it would have been likely that this and other health outcomes would have shown significant improvements, as was seen in depression (which was studied on n=259 patients), rather than trends. It is the investigators intention to add results to the body of research from a future full-scale trial.

Currently Mindfulness-based treatment is creating lively research interest. Two recent systematic reviews report positive effects on somatisation disorders and psychological stress. Although there is no ongoing study on patients with CPP, other chronic diseases with strong psychological components of depression and anxiety such as COPD and the RFPB-funded pilot study PATHWAYS on Pulmonary Arterial Hypertension are underway.

Of particular interest, due to the similarities in study design to MEMPHIS, is a recently closed pilot study, MIMS (UKCRN ID 13105) that investigated adjustment to multiple sclerosis.

In MIMS meditation teaching was delivered by videoconference. Web-based delivery has also been explored and shown to be feasible for reducing stress, anxiety and depression; both options are lacking the flexibility of a smartphone app, which is being proposed. There is evolving work on care pathways through primary secondary and tertiary levels for patients with CPP and recently mindfulness meditation has been introduced in Dorset, albeit delivered face-to-face. This could be replaced by cheaper and more flexible app-delivered meditation training.

This study will address the knowledge gaps and provide by:

1. Providing feasibility data for a large multicentre RCT aimed at rigorously testing Mindfulness meditation in CPP
2. Establishing whether this app could be seamlessly integrated into CPP pathways

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of organic and non-organic chronic pelvic pain (CPP) for six months or more
* Age ≥ 18 years
* Be capable of understanding the information provided, with use of an interpreter if required and being able to understand simple English as is used in the app

Exclusion Criteria:

* Males
* Absence of diagnosis of organic and non-organic chronic pelvic pain (CPP)
* Diagnosis of organic and non-organic chronic pelvic pain (CPP) lasting for less than 3 months
* Age < 18 years
* No access to a Personal computer or smart phone
* Unable to speak / understand English
* Current users of the app content available to the public

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Duration of recruitment | 6 months
  Length of time it will take to recruit 90 participant from the time recruitment starts
Patient adherence to app use | first 8 weeks post-randomisation

SECONDARY OUTCOMES:
Quality of life score-Physical Functioning subscale (as measured by the RAND Short form Health Survey (SF-36) | at 60 days, 3 months, and 6 months post-randomisation
Quality of life score-Social Functioning subscale (as measured by the RAND Short form Health Survey (SF-36) | at 60 days, 3 months, and 6 months post-randomisation
Quality of life score-Pain subscale (as measured by the RAND Short form Health Survey (SF-36) | at 60 days, 3 months, and 6 months post-randomisation
Quality of life score-General Health subscale (as measured by the RAND Short form Health Survey (SF-36) | at 60 days, 3 months, and 6 months post-randomisation
Depression score as measured by the Hospital Anxiety and Depression Scale (HADS) | at 60 days, 3 months, and 6 months post-randomisation
Anxiety score (as measured by HADS) | at 60 days, 3 months, and 6 months post-randomisation
Mindfulness score as measure by the Cognitive and Mindfulness - Revised (CAMS - R) scale | at 60 days, 3 months, and 6 months post-randomisation
Pain related disability score (as measured by the Chronic Pain Grade (CPG) disability subscale | at 60 days, 3 months, and 6 months post-randomisation
Self efficacy score (as measured by the Pain Self-Efficacy Questionnaire (PSEQ) | at 60 days, 3 months, and 6 months post-randomisation
Pain acceptance score (as measured Chronic Pain Acceptance Questionnaire (CPAQ-8) | at 60 days, 3 months, and 6 months post-randomisation
Sexual Health Outcomes score (as measured by Sexual Health Outcomes in Women Questionnaire (SHOW-Q) | at 60 days, 3 months, and 6 months post-randomisation
Subjective outcome score (as measured by Measure Yourself Medical Outcome Profile (MYMOP) | at 60 days, 3 months, and 6 months post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ball, PhD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is a feasibility study. data will be used to inform design of a full-scale trial.

REFERENCES:
- [Derived] Forbes G, Newton S, Cantalapiedra Calvete C, Birch J, Dodds J, Steed L, Rivas C, Khan K, Rohricht F, Taylor S, Kahan BC, Ball E. MEMPHIS: a smartphone app using psychological approaches for women with chronic pelvic pain presenting to gynaecology clinics: a randomised feasibility trial. BMJ Open. 2020 Mar 12;10(3):e030164. doi: 10.1136/bmjopen-2019-030164. PMID 32165549
- [Derived] Ball E, Newton S, Kahan BC, Forbes G, Wright N, Cantalapiedra Calvete C, Gibson HAL, Rogozinska E, Rivas C, Taylor SJC, Birch J, Dodds J. Smartphone App Using Mindfulness Meditation for Women With Chronic Pelvic Pain (MEMPHIS): Protocol for a Randomized Feasibility Trial. JMIR Res Protoc. 2018 Jan 15;7(1):e8. doi: 10.2196/resprot.7720. PMID 29335232